CLINICAL TRIAL: NCT01482754
Title: Rapid Rituximab Infusion at 90-minute Among Non-Hodgkin Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Prof. Chng Wee Joo, National University Hospital, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB Ref. 2011/02052
Record Dates: First submitted 2011-11-28; First posted 2011-12-01 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab Infusion at 90-minutes (Experimental)
  Interventions: Drug: Rituximab (Mabthera®, Roche Pty Ltd, Basel, Switzerland)

INTERVENTIONS:
Drug: Rituximab (Mabthera®, Roche Pty Ltd, Basel, Switzerland) — Recommended and approved dosage of Rituximab is 375mg/m2. The recommended guideline for Rituximab infusion for first cycle is commencing at an infusion rate of 50mg/hr for the first 30 minutes. If tolerated well, the subsequent increments will step up to 50mg/hr every 30 minutes to a maximum dose of 400mg/hr. For second and subsequent infusions, the infusion rate commences at 100mg/hr with 30 minute increments of 100mg/hr to a maximum dose of 400mg/hr. The first and subsequent infusion generally completes between 5-6 and 3-4 hours respectively.

SUMMARY:
This is an observational prospective cohort study design to evaluate the safety of rapid Rituximab infusion at 90 minutes for Non-Hodgkin Lymphoma (NHL) patients. The secondary aim is to measure the number of rejected chemotherapy administration on schedule. Non-Hodgkin lymphoma patients who tolerated well for at least 2 cycles of standard infusion of Rituximab without grade 3 or 4 adverse events will be recruited in the study. In this study, the first 20% of the total dose of rituximab will be administered over 30 minutes. When subjects tolerate the infusion and stable vital signs, the remaining 80% of the total dose will be administered over 60 minutes. Prior administration of Rituximab, premedication will be given to the subjects including PO Paracetamol 1g, IV Diphenhydramine 25/50mg and/or IV Hydrocortisone 100mg. The duration of subjects involvement in the study approximately takes 72 hours. Adverse events that occur within the first 24 hours of infusion will be evaluated if related to Rituximab infusion as some subjects are receiving combination chemotherapy with rituximab. This study will recruit both in patients and out-patients. A phone call to monitor subject's health will be made post 24, 48, 72 hours of rituximab infusion. The findings from this study will add evidence to the safety of rapid Rituximab infusion at 90 minutes. If the outcome is favourable, NUH will consider adopting the new infusion rate for Rituximab infusion for patients who tolerated at least 2 cycles of standard infusion recommended by the drug manufacturer.

The study hypothesizes that rapid Rituximab infusion at 90 minutes is safe for NHL patients.

DETAILED DESCRIPTION:
The recommended guideline for Rituximab infusion for first cycle is to be commencing at an infusion rate of 50mg/hr for the first 30 minutes. If tolerated well, subsequent increments will step up to 50mg/hr every 30 minutes to a maximum dose of 400mg/hr. For second and subsequent infusions, the infusion rate commences at 100mg/hr with 30 minute increments of 100mg/hr to a maximum dose of 400mg/hr. The first and subsequent infusion generally completes between 5-6 and 3-4 hours respectively.

Lengthy infusions translate into higher costs and longer waiting times for patients due to scant resources. Therefore, there is growing interest globally in shortening the overall infusion times to either 90 or 60-minutes. A recent systematic review evaluating safety of rapid Rituximab infusion has confirmed that Rituximab at 90-minutes is safe for NHL patients. However 60-minute infusion was not recommended for neither NHL nor chronic lymphocytic leukemia (CLL) patients due to lack of evidence.

Although the rapid Rituximab infusion at 90-minute has been tested among Singapore population in National Cancer Centre, it was not being evaluated among the cohort of patients who received treatment in National University Hospital Singapore. As rapid Rituximab infusion remain off label use, this research study intend to evaluate the safety of rapid Rituximab infusion at 90-minute among NHL patients.

The selected doses will be 375mg/m2 as recommended and approved by FDA.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of NHL is confirmed through histology report.
* Adult with age 21 years old and above
* Tolerated first and second cycles or at least two cycles of Rituximab infusion at recommended rate without Grade 3 or 4 adverse event during infusion
* Presence of any co-morbidity
* Ability to provide informed consent

Exclusion Criteria:

Subjects who diagnosed with NHL with high lymphocytes counts will be excluded from the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety of rapid Rituximab infusion at 90-minute for NHL | 72 hours
  This is an observational prospective cohort study design with single group. The duration of subjects involvement in the study is approximately 72 hours. Adverse events that will occur within first 24 hours of infusion will be evaluated if related to Rituximab infusion as some subjects are receiving combination chemotherapy with rituximab. This study will recruit both in-patients and out-patient. A phone call to monitor subject's health will be made post 24, 48 and 72 hours of rituximab infusion.

SECONDARY OUTCOMES:
number of rejected chemotherapy administration on schedule. | 5-6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Chng Wee Joo, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore